CLINICAL TRIAL: NCT06152835
Title: The BuKoBc Project: Building a Deeper Knowledge on Breast Milk Composition
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Medical Doctor, PhD, Professor, Federico II University
Other Study IDs: 14/2023
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Breastfeeding Italian women: Italian women, aged 20-40 years who breastfeed children born at full term
  Interventions: Other: Data and breast milk samples collection

INTERVENTIONS:
Other: Data and breast milk samples collection — Breast milk samples and, clinical, anamnestic and lifestyle data collection

SUMMARY:
Breast milk is considered the gold standard for infant nutrition thanks to its ability to provide adequate nutrition and a high amount of protective factors for the baby's health. According to the guidelines of the World Health Organization (WHO), exclusive feeding with breast milk should be conducted until the end of 6 months of life and should be continued in the following months with the simultaneous introduction of complementary foods. Several evidence demonstrates that breast milk intake is associated with positive health outcomes, both during infancy and later in the life. Given the protective role of breast milk for the health of the child and the future adult, studying its content is of fundamental importance to have an integrated vision of the biological effects of its components on the child health, and of the factors that are able to modulate its composition. The "Building a Deeper Knowledge on Breast Milk Composition" (BuKoBc) project was designed to study the content of human milk in its entirety and at different times during the feeding and day, also in relation to environmental factors capable of modulating its composition. The results of this study may provide data on optimal reference ranges for nutrient intake in breastfed infants and may provide guidance for defining optimal nutrient intake for infants who cannot be breastfed. Furthermore, the in-depth study of the environmental factors capable of influencing the composition of breast milk will allow the development of nutritional intervention strategies for the breastfeeding mother in order to positively modulate the composition of her milk.

ELIGIBILITY:
Inclusion Criteria:

* Italian women aged between 20 and 40 years who exclusively breastfeed children born at term from normal pregnancy
* Written informed consent

Exclusion Criteria:

* Non-Italian women;
* Age <20 and >40 years;
* Mothers of children born preterm;
* Non-exclusive breastfeeding;
* Mothers suffering from chronic diseases:
* malignancies;
* immunodeficiencies;
* chronic infections;
* autoimmune diseases;
* chronic inflammatory intestinal diseases;
* celiac disease;
* genetic-metabolic diseases;
* cystic fibrosis;
* chronic lung diseases;
* malformations of the cardiovascular/respiratory/gastrointestinal system;
* neuropsychiatric disorders;
* neurological diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 Italian women, aged 20-40 years, who breastfed children born at full term, observed at the specialist pediatric clinics of the "Federico II" University Hospital of Naples, of the "La Sapienza University of Rome", of the "La Statale University of Milan", the "University of Pisa" and the "University of Verona".
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
To analyze the contents of breast milk completely and at different times during the feeding and during the day. | 36 months
  6 milk samples of at least 5 ml each will be collected at the beginning and end of the morning feeding, at the beginning and end of the afternoon feeding, and at the beginning and end of the evening feeding.
Nutritional composition analysis (macro and micronutrients) | 36 months
  Mass spectrometry analyzes will be performed.
Metagenomic analysis | 36 months
  Shotgun analysis will be performed.
Metabolomics analysis | 36 months
  Mass spectrometry analyzes will be performed.
MicroRNA analysis | 36 months
  TaqMan MicroRNA Assays will be adopted.
Compounds derived from ultraprocessed foods and from packaging analyses | 36 months
  Mass spectrometry analyzes will be performed.

SECONDARY OUTCOMES:
To analyze the environmental factors capable of modulating the composition of breast milk | 36 months
  Maternal energy and nutrient intake, maternal ultra-processed food intake, level of adherence to the Mediterranean Diet, nutritional status, body composition, lifestyle, level of physical activity, level of education, intake of medications, food supplements, prebiotics, probiotics and synbiotics, consumption of alcohol, caffeine and tobacco will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No